CLINICAL TRIAL: NCT00438451
Title: A Multicentre, Double-blind, Randomized, Phase IV Clinical Trial Comparing the Safety, Tolerability and Efficacy of Levetiracetam Versus Lamotrigine and Carbamazepine in the Oral Antiepileptic Therapy of Newly Diagnosed Elderly Patients With Focal Epilepsy.
Brief Title: Study on the Treatment of Elderly Patients With Older and Newer Antiepileptic Drugs
Acronym: STEP-ONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: UCB Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Konrad J. Werhahn, Prof of Neurology, Head Section on Epilepsy, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STEPONE05; ISRCTN: 94839639; EudraCT Number:2005-003324-19
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-01

CONDITIONS: Focal Epilepsy
Keywords: elderly; focal epilepsy; anticonvulsive; treatment; levetiracetam; lamotrigine; carbamazepine
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam; Carbamazepine; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levetiracetam (Active Comparator): Levetiracetam
  Interventions: Drug: Levetiracetam
- Carbamazepine (Active Comparator): Carbamazepine
  Interventions: Drug: Carbamazepine
- Lamotrigine (Active Comparator): Lamotrigine
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Levetiracetam — LEV 250 mg capusles: week 1 and 2 0-0-1, week 3 and 4 1-0-1, week 5: 1-0-2, week 6: 2-0-2. Patients may take 2 to 12 per day (500 - 3000 mg)during maintenance.
  Arms: Levetiracetam
Drug: Carbamazepine — CBZ 100 mg capusles: week 1 and 2: 0-0-1, week 3 and 4: 1-0-1, week 5: 1-0-2, week 6: 2-0-2. Patients may take 2 to 12 per day (200 - 1200 mg) during maintenance depending on tolerance and efficacy.
  Arms: Carbamazepine
Drug: Lamotrigine — LTG 25 mg encapsulated: week 1 and 2: 0-0-1, week 3 and 4: 1-0-1, week 5: 1-0-2, week 6: 2-0-2. Patients may take 2 to 12 caps. per day (50 - 300 mg)during maintenance depending on tolerance and efficacy.
  Arms: Lamotrigine

SUMMARY:
In this clinical trial patients with newly diagnosed focal epilepsy aged 60 years or older receive three different antiepileptic drugs in a double-blind, randomized design over a period of 58 weeks. All drugs are licensed for the treatment of epilepsy. The primary endpoint of this study will be retention rate at 58-weeks, since it reflects both efficacy and tolerability.

DETAILED DESCRIPTION:
Indication: Focal Epilepsy Objectives: To evaluate the tolerability and efficacy of levetiracetam (LEV) in newly diagnosed elderly patients (aged 60 yrs or above) with focal epilepsy compared to lamotrigine (LTG) or carbamazepine slow release (CBZ).

Primary Outcome: The primary outcome will be the 58-week retention rate measured by the number of drop outs due to adverse events or seizures from day 1 of treatment.

Secondary Outcome: Proportion of patients remaining seizure-free at week 30 (Visit 4); proportion of patients remaining seizure free at week 58 (Visit 6); the time (in days) to first break-through seizure (from day 1 of treatment); the absolute seizure frequency during the maintenance (over 52 weeks) phase; proportion of seizure-free days during the maintenance phase for subjects who enter the maintenance phase; the frequency of adverse events (from day 1 of treatment); QOLIE-31 results at V6; Portland Neurotoxicity scale at V6; results of cognitive testing (EpiTrack© by UCB).

Trial Design: This is a randomized, double-blind, multicenter Phase IV study using a parallel group design with three treatment groups. The study will consist of a 6-week titration-phase and a 52-week maintenance phase. Patients who successfully complete the trial (final visit, V6) will be unblinded and offered either to continue on their current drug or be changed to an alternative antiepileptic drug (AED) treatment of choice.

Population: Patients aged 60 years or above with new onset focal epilepsy i.e. either at least one epileptic seizure in the last 6 months and focal epileptiform discharges on EEG or a relevant lesion on CT/MRI or a total of 2 epileptic seizures, one of which occurring in the last 6 months prior inclusion. Patients with acute (< 2 weeks) symptomatic epileptic seizures due to acute brain abnormalities (i.e. haemorrhage or cerebral infarct), or contraindications against any of the drugs in trial will be excluded.

Sample Size: 360 patients to be included, 120 patients per treatment arm. Investigational Medicinal Product(s): Levetiracetam, lamotrigine, carbamazepine-slow release Trial Duration and Dates: Duration of treatment: 6 weeks titration phase, 52 weeks maintenance phase.

Follow up: At the end of trial subjects will be unblinded and may choose to continue on the medication or taper the trial medication and be treated with an alternative drug at the investigators discretion. The patient will receive a dosing schedule and a referral letter for his/her physician.

Duration of trial: approximately 2 years. Start of recruitment: January 2007 Projected number of centres: 75 Number of countries: 3 (Germany, Switzerland, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 yrs or above.
* New onset focal epilepsy i.e. either at least one epileptic seizure in the last 6 months and focal epileptiform discharges on EEG or a relevant lesion on CT/MRI or at least 2 epileptic seizures, one of which occurring in the last 6 months prior inclusion.
* No previous AED treatment, except for a period not longer than 4 weeks prior to inclusion (V0).
* Ability of subject to understand verbal and written instructions, to comply with all study requirements, and to comprehend character and individual consequences of the clinical trial.
* Written informed consent before enrolment in the trial.

Exclusion Criteria:

* Acute symptomatic epileptic seizures occurring acutely within a 2 week period after the onset of an acute illness such as cerebral haemorrhage, cerebral infarct, rapid progressive malignancy or other acute brain abnormalities (i.e. encephalitis, hypoxic brain damage, trauma, metabolic derangement, following brain surgery).
* Dementia (as defined by history)
* Renal insufficiency as defined by GFR < 50 mL/min.
* Increased liver enzymes (GOT, GPT, gGT) or increased bilirubin ≥ 2-fold the upper limit of normal (ULN).
* Pre-treatment with valproic acid within the four weeks prior inclusion (V0).
* Contraindication against or history of hypersensitivity to any of the investigational medicinal products or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal products.
* Participation in other clinical trials and observation period of competing trials within the last 2 months, respectively.
* History of drug or alcohol abuse within the last 2 years.
* Medical condition which interferes with the participation in the trial according to the opinion of the investigator.
* Patients with life expectancy < 1 year due to malignant disease
* Psychiatric morbidity requiring legal guardianship.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2007-01; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konrad J Werhahn, MD, Study Chair — Johannes Gutenberg University, Department od Neurology; Günter Kraemer, MD, Study Director — Swiss Epilepy Centre; Eugen Trinka, MD, Study Director — Medical University of Salzburg, Department of Neurology, Austria
Locations (1):
- Department of Neurology, University of Mainz Medical Centre, Mainz, Germany

REFERENCES:
- [Background] Rowan AJ, Ramsay RE, Collins JF, Pryor F, Boardman KD, Uthman BM, Spitz M, Frederick T, Towne A, Carter GS, Marks W, Felicetta J, Tomyanovich ML; VA Cooperative Study 428 Group. New onset geriatric epilepsy: a randomized study of gabapentin, lamotrigine, and carbamazepine. Neurology. 2005 Jun 14;64(11):1868-73. doi: 10.1212/01.WNL.0000167384.68207.3E. PMID 15955935
- [Background] Brodie MJ, Chadwick DW, Anhut H, Otte A, Messmer SL, Maton S, Sauermann W, Murray G, Garofalo EA; Gabapentin Study Group 945-212. Gabapentin versus lamotrigine monotherapy: a double-blind comparison in newly diagnosed epilepsy. Epilepsia. 2002 Sep;43(9):993-1000. doi: 10.1046/j.1528-1157.2002.45401.x. PMID 12199724
- [Derived] Werhahn KJ, Trinka E, Dobesberger J, Unterberger I, Baum P, Deckert-Schmitz M, Kniess T, Schmitz B, Bernedo V, Ruckes C, Ehrlich A, Kramer G. A randomized, double-blind comparison of antiepileptic drug treatment in the elderly with new-onset focal epilepsy. Epilepsia. 2015 Mar;56(3):450-9. doi: 10.1111/epi.12926. Epub 2015 Feb 12. PMID 25684224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 study centres in three countries participated in this study (31 in Germany, 5 in Austria, 7 in Switzerland). The number of patients recruited in each country (242 Germany, 55 Austria, 29 Switzerland) and per centre (range from 1 to 53) was heterogeneous.
  Therefore, centre effects were explored by pooling the centres with less than 20 subjects.
Pre-assignment Details: In total, 361 patients were randomized. 359 patients were analysed ITT (patient 0213 did not suffer from epilepsy, patient 3604 should not have been asked for informed consent, because of his legal guardianship).
Groups:
- Levetiracetam: Levetiracetam 250mg: capsules, each containing one Levetiracetam 250mg film-coated tablet.
  During titration phase, subjects received 1 capsule in the evening in the first 14 days, 2 capsules (1 in the morning and 1 in the evening) in week 3 and 4, 3 capsules in week 5 (1 in the morning and 2 in the evening) and 4 capsules from week 6 onwards (2 in the morning and 2 in the evening). During maintenance phase, dose adjustments could be made according to tolerability and seizure control in steps of 1 capsule per week. Dosages between 2 to 12 capsules per day were allowed.
- Carbamazepine: Carbamazepine 100mg: capsules, each containing half of one Carbamazepine 200mg slow release tablet.
  During titration phase, subjects received 1 capsule in the evening in the first 14 days, 2 capsules (1 in the morning and 1 in the evening) in week 3 and 4, 3 capsules in week 5 (1 in the morning and 2 in the evening) and 4 capsules from week 6 onwards (2 in the morning and 2 in the evening). During maintenance phase, dose adjustments could be made according to tolerability and seizure control in steps of 1 capsule per week. Dosages between 2 to 12 capsules per day were allowed.
- Lamotrigine: Lamotrigine 25mg: capsules, each containing one Lamotrigine 25mg tablet. During titration phase, subjects received 1 capsule in the evening in the first 14 days, 2 capsules (1 in the morning and 1 in the evening) in week 3 and 4, 3 capsules in week 5 (1 in the morning and 2 in the evening) and 4 capsules from week 6 onwards (2 in the morning and 2 in the evening). During maintenance phase, dose adjustments could be made according to tolerability and seizure control in steps of 1 capsule per week. Dosages between 2 to 12 capsules per day were allowed.
Period: Overall Study
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Started | 122 | 121 | 118
Safety Population | 122 | 121 | 117
ITT Population | 122 | 120 | 117
Maintenance Phase (Week 7-58) | 93 | 89 | 93
Completed | 75 | 55 | 65
Not Completed | 47 | 66 | 53

BASELINE CHARACTERISTICS:
Groups:
- Levetiracetam: Levetiracetam 250mg
- Carbamazepine: Carbamazepine 100mg
- Lamotrigine: Lamotrigine 25mg
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine | Total
Number analyzed (Participants) | 122 | 120 | 117 | 359
Age Continuous [Mean (Standard Deviation); unit: years] — Age is shown for ITT population
  years | 71.8 (7.49) | 71.7 (6.66) | 70.7 (7.43) | 71.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender is shown for ITT population
  Participants
    Female | 41 | 55 | 48 | 144
    Male | 81 | 65 | 69 | 215
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race is shown for ITT population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 122 | 120 | 117 | 359
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Region of enrollment is shown for ITT population
  participants
    Germany | 95 | 92 | 91 | 278
    Austria | 18 | 18 | 16 | 52
    Switzerland | 9 | 10 | 10 | 29
Epilepsy history - number of seizures [Mean (Standard Deviation); unit: number of seizures] — is shown for ITT population
  number of seizures | 3.8 (9.85) | 4.8 (10.78) | 2.7 (3.14) | 3.75 (8.69)
Epilepsy history - Aura [Number; unit: participants] — is shown for ITT population "NA" refer to the fact that the epilepsy history - Aura is unknown
  participants
    Yes | 23 | 28 | 21 | 72
    No | 99 | 92 | 95 | 286
    NA | 0 | 0 | 1 | 1
Epilepsy history - Autonomic seizure [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 1 | 2 | 0 | 3
    No | 121 | 118 | 117 | 356
Epilepsy history - Dialeptic seizure [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 13 | 15 | 18 | 46
    No | 109 | 105 | 99 | 313
Epilepsy history - Motor seizure [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 95 | 101 | 95 | 291
    No | 27 | 19 | 22 | 68
Epileptic history - Special seizure [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 8 | 13 | 12 | 33
    No | 114 | 107 | 105 | 326
EEG (electroencephalogram) pathological [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 86 | 84 | 71 | 241
    No | 35 | 36 | 45 | 116
    Missing | 1 | 0 | 1 | 2
MRT (Magnetic Resonance Tomograhy) pathological [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 59 | 63 | 62 | 184
    No | 11 | 10 | 13 | 34
    Missing | 52 | 47 | 42 | 141
CCT (Cranial Computed Tomography) pathological [Number; unit: participants] — is shown for ITT population
  participants
    Yes | 76 | 82 | 64 | 222
    No | 23 | 19 | 19 | 61
    Missing | 23 | 19 | 34 | 76

OUTCOME MEASURES:

1. Primary Outcome: 58-week Retention Rate Measured by the Number of Drop Outs Due to Adverse Events or Seizures From Day 1 of Treatment
Time Frame: 58 weeks
Population: ITT population:
  All randomized patients were included in the Intention-to-Treat (ITT) population except patients that were not evaluable for efficacy e.g. patients without epilepsy or patients not able to comply with the study requirements.
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 122 | 120 | 117
proportion of participants | 0.61 [0.53 to 0.70] | 0.46 [0.37 to 0.55] | 0.56 [0.47 to 0.65]
Statistical Analysis 1: Comparison: Levetiracetam vs Carbamazepine; Test type: Superiority or Other; p = 0.0201, Fisher Exact
Statistical Analysis 2: Comparison: Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.1536, Fisher Exact
Statistical Analysis 3: Comparison: Levetiracetam vs Lamotrigine; Test type: Superiority or Other; p = 0.3615, Fisher Exact
Statistical Analysis 4: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.0478, Fisher Exact
Statistical Analysis 5: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.0578, Regression, Logistic; adjusted for treatment (p=0.0578), country (p=0.4649), pooled sites (p=0.4420) and number of concurrent diseases (p=0.0192); Odds Ratio (OR) = 1.838, 95% CI 2-sided [1.092 to 3.093] — Odds ratio given here is for comparison "LEV vs CBZ": OR=1.838 KI=(1.092-3.093) "LEV vs LTG": OR=1.169 KI=(0.689-1.984) "CBZ vs LTG": OR=0.636 KI=(0.377-1.073) "Number of concurrent diseases": OR=0.921 KI=(0.859-0.987)

2. Secondary Outcome: Time to Drop Out
Description: number of days between randomization and premature discontinuation of the study
Time Frame: 58 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 122 | 120 | 117
days | NA [NA to NA] — less than 50% of patients dropped out | 265 [119 to NA] — not enough patients dropped out | NA [270 to NA] — less than 50% of patients dropped out
Statistical Analysis 1: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.0596, Log Rank

3. Secondary Outcome: Percentage of Patients Remaining Seizure-free at Week 30 (Visit 4)
Description: Percentage of patients experiencing no seizures until week 30 (Visit 4) and did not discontinue the study until week 30.
Time Frame: Week 30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 122 | 120 | 117
percentage of participants | 48 | 39 | 49
Statistical Analysis 1: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.2517, Fisher Exact

4. Secondary Outcome: Percentage of Patients Remaining Seizure Free at Week 58 (Visit 6)
Description: Percentage of patients experiencing no seizures until week 58 (Visit 6) and did not discontinue the study until week 58.
Time Frame: week 58
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 122 | 120 | 117
percentage of participants | 43 | 33 | 38
Statistical Analysis 1: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.3303, Fisher Exact

5. Secondary Outcome: The Time (in Days) to First Break-through Seizure (From Day 1 of Treatment)
Time Frame: over the whole duration of 58 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 122 | 120 | 117
days | NA [NA to NA] — could not be estimated since there were less than 50% events | NA [NA to NA] — could not be estimated since there were less than 50% events | NA [308 to NA] — could not be estimated since there were less than 50% events
Statistical Analysis 1: Comparison: Levetiracetam vs Carbamazepine vs Lamotrigine; Test type: Superiority or Other; p = 0.5022, Log Rank

6. Secondary Outcome: The Absolute Seizure Frequency During the Maintenance Phase (Weeks 7 - 58)
Description: Seizure frequency was assessed by investigators in the CRF at the Visits V3, V4, V5 and V6.
  The absolute seizure frequency during the maintenance phase was defined as the sum of those entries.
Time Frame: over 52 weeks
Population: Completer population:
  The completer population comprises all patients still being in the study at week 58 (This definition deviates minimally from the protocol. It could not be assessed from the CRF data, if patients were on treatment).
Measure: Number; unit: number of seizures
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 75 | 55 | 65
number of seizures | 168 | 131 | 130

7. Secondary Outcome: Proportion of Seizure-free Days During the Maintenance Phase for Subjects Who Enter the Maintenance Phase
Time Frame: 52 weeks
Population: Patients of ITT population who reached the maintenance phase
Measure: Number; unit: proportion of seizure-free days
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 91 | 87 | 91
proportion of seizure-free days | 0.99 | 0.99 | 0.99

8. Secondary Outcome: QOLIE-31 (Quality Of Life In Epilepsy) Results at V6
Description: The QOLIE-31 is a 31 item score that measures the quality of life in epilepsy (each item with a range of 0 to 100). There are 7 sub-scores seizure worry (items 11,21,22,23,25), overall quality of life (items 1,14), emotional well-being (items 3,4,5,7,9), energy/fatigue (items 2,6,8,10), cognitive functioning (items 12,15,16,17,18,26), medication effects (items 24,29,30) and social functioning (13,19,20,27,28). These scores were combined to a total score by Total score = seizure worry*0.08 + overall quality of life*0.14 + emotional well-being*0.15 + energy/fatigue*0.12 + cognitive functioning*0.27 + medication effects*0.03 + social functioning*0.21 For all scores, higher values indicate better quality of life. Each score has a possible range from 0 to 100.
Time Frame: 58 weeks, final visit
Population: Patients of ITT population who filled out QOLIE-31 at V6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 90 | 90 | 89
units on a scale
  Seizure worry | 85.1 (19.89) [25 to 100] | 75.4 (26.87) [0 to 100] | 75.0 (26.26) [0 to 100]
  Overall quality of life | 67.2 (21.76) [10 to 100] | 65.0 (20.65) [5 to 100] | 67.1 (20.96) [10 to 100]
  Emotional well-being | 72.0 (19.42) [16 to 100] | 69.8 (18.76) [20 to 100] | 67.4 (20.25) [16 to 100]
  Energy/fatigue | 60.8 (21.03) [15 to 100] | 54.5 (21.33) [5 to 95] | 59.8 (22.07) [10 to 100]
  Cognitive functioning | 75.1 (19.48) [10 to 100] | 68.9 (20.96) [18 to 100] | 68.0 (21.11) [10 to 100]
  Medication effects | 77.6 (26.78) [0 to 100] | 70.6 (28.21) [0 to 100] | 72.6 (30.34) [0 to 100]
  Social functioning | 81.1 (19.23) [25 to 100] | 76.3 (25.49) [5 to 100] | 76.7 (24.28) [5 to 100]
  Total Score | 73.9 (15.89) [26 to 100] | 68.9 (17.80) [30 to 96] | 69.1 (17.12) [17 to 96]
  Health Scale | 69.5 (19.28) [20 to 100] | 65.7 (21.21) [10 to 100] | 67.5 (19.84) [20 to 100]

9. Secondary Outcome: Portland Neurotoxicity Scale (PNS) at V6
Description: The PNS is a 15-item scale. Each item can be scored from 1 to 9. There are a total score (includes all items, range:15 to 135) and two subscores: The cognitive toxicity subscore (10 items: Energy Level, Memory, Interest, Concentration, Forgetfulness, Sleepliness, Moodiness, Alertness, Attention Span, Motivation, range:10 to 90) and the somatomoto subscore (5 items: Vision, Walking, Coordination, Tremor, Speech, range:5-45). The score is calculated by taking the mean of all non-missing values times the number of items.
  Lower values indicate better quality of life.
Time Frame: at week 58
Population: Patients of ITT population who filled out PNS at V6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 90 | 90 | 89
units on a scale
  Cognitive toxicity subscore | 22.2 (12.52) [10 to 79] | 27.3 (15.71) [10 to 82] | 23.7 (11.44) [10 to 66]
  Somatomotor subscore | 10.5 (5.53) [5 to 28] | 11.4 (6.96) [5 to 35] | 10.8 (5.42) [5 to 31]
  Total Score | 32.7 (16.81) [15 to 107] | 38.7 (21.73) [15 to 110] | 34.5 (15.67) [15 to 83]

10. Secondary Outcome: Results of Cognitive Testing (EpiTrack© by UCB) - Score at V6
Description: EPITrack-Score shows the performance of attention and executive functions. Higher values indicate a better performance. The results of EPITrack Score ranges between 7 and 45.
Time Frame: week 58
Population: Patients of ITT population who had data at V6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 84 | 84 | 85
units on a scale | 26.0 (7.22) [11 to 38] | 26.0 (7.05) [8 to 39] | 25.4 (6.82) [7 to 39]

11. Secondary Outcome: Results of Cognitive Testing (EpiTrack© by UCB) - Categories at V6
Description: Evaluation of current testing at V6:
  ≥29 score points: Inconspicuous; 26 to 28 score points: Borderline;
  ≤25 score points: Impaired
Time Frame: 58 weeks
Population: Patients of ITT population with data at V6
Measure: Number; unit: participants
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 84 | 84 | 85
participants
  Without pathological findings | 38 | 34 | 31
  Borderline | 10 | 17 | 15
  Impaired | 36 | 33 | 39

12. Secondary Outcome: Results of Cognitive Testing (EpiTrack© by UCB) - Changes to Baseline (V0) at Week 58 (V6)
Description: Evaluation of Changes
  Changes in the EpiTrack® Score were categorized as follows:
  ≥5 score points: Improved;
  -3 to 4 score points: Unchanged;
  ≤-4 score points: Worsened
Time Frame: week 58
Population: Patients of ITT population with data at V6 and V0
Measure: Number; unit: participants
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Number analyzed (Participants) | 82 | 80 | 81
participants
  Improved | 15 | 16 | 15
  Unchanged | 61 | 56 | 53
  Worsened | 6 | 8 | 13

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from day 1 of treatment
Arm/Group | Levetiracetam | Carbamazepine | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 33/122 | 36/121 | 32/117
Other Adverse Events (participants affected / at risk) | 108/122 | 108/121 | 110/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=122) | Carbamazepine (N=121) | Lamotrigine (N=117)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute mycardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthroscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amnestic disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 5 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Suicidal behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bursa removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Meningioma surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=122) | Carbamazepine (N=121) | Lamotrigine (N=117)
Constipation (Gastrointestinal disorders) | 2 (2) | 15 (16) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 13 (14) | 14 (17)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 7 (8)
Nausea (Gastrointestinal disorders) | 11 (15) | 18 (21) | 17 (23)
Vomiting (Gastrointestinal disorders) | 5 (10) | 6 (11) | 7 (7)
Fatigue (General disorders) | 31 (48) | 46 (51) | 23 (29)
Gait disturbance (General disorders) | 8 (8) | 10 (11) | 5 (6)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 7 (7)
Nasopharyngitis (Infections and infestations) | 20 (26) | 13 (18) | 8 (10)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (7) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 18 (20) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (4) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 7 (12)
Convulsion (Nervous system disorders) | 5 (5) | 7 (9) | 11 (23)
Dizziness (Nervous system disorders) | 35 (52) | 31 (35) | 36 (44)
Epilepsy (Nervous system disorders) | 19 (35) | 11 (16) | 14 (22)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 7 (14)
Headache (Nervous system disorders) | 31 (46) | 29 (39) | 29 (44)
Memory impairment (Nervous system disorders) | 5 (6) | 7 (7) | 5 (6)
Partial seizures (Nervous system disorders) | 1 (3) | 5 (19) | 8 (10)
Tremor (Nervous system disorders) | 6 (6) | 5 (6) | 6 (10)
Depression (Psychiatric disorders) | 4 (5) | 6 (6) | 4 (4)
Sleep disorder (Nervous system disorders) | 4 (5) | 5 (5) | 9 (10)
Renal failure (Renal and urinary disorders) | 9 (9) | 0 (0) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 9 (9) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study was supported (as investigator-initated trial) by an educational grant from UCB GmbH, Germany. A disclosure restriction applies on the PI in that UCB can review results communications prior to public release and can embargo communications regarding trial results for a period of 90 days from the time submitted. As of Jan-01-2012 the study chair is an employee to UCB Biosciences GmbH working as Medical Director in the Therapeutic Area CNS within Global Projects and Development.